CLINICAL TRIAL: NCT01038856
Title: Phase II Trial of Erlotinib in Patients With JAK-2 V617F Positive Polycythemia Vera
Brief Title: Trial of Erlotinib in Patients With JAK-2 V617F Positive Polycythemia Vera
Acronym: OSI-TAR-766
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the sponsor
Sponsor: University of Oklahoma (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2249
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- +JAK2V61F mutation (Experimental): Patients with MPN diagnoses and polycythemia vera who also have a confirmed JAK2V617F mutation
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib supplied as tablets; oral dose of erlotinib of 150 mg daily to be continued for 16 weeks. Responders will continue for up to 12 months, non-responders will cease taking erlotinib
  Other Names: Tarceva; OSI-744

SUMMARY:
The primary objective of this study is to determine the overall response rate to erlotinib in patients with polycythemia vera (PV). Response rate will be assessed by improvement in the complete blood count, ultrasound of the spleen, and JAK2 molecular status. It is purposed in this study to explore a possible molecular targeting of the driving mechanism of PV.

DETAILED DESCRIPTION:
This is a phase II open-label study. Patients will be screened for MPN diagnoses and patients with Polycythemia vera proven to have JAK2V617F mutation will be given the option to enroll. Consenting patients will take erlotinib daily for 16 weeks. Blood work and pharmacokinetics will be drawn for serum level monitoring. Doses will be administered according to side effects or held. First assessment will be at day 15 wth subsequent assessments at 28 day intervals. Non-responders will be taken off the study and managed according to standard of care. Patients who do respond will continue taking the therapy for a total of 12 months. Observation will be for a total of 12 months after finishing treatment. In addition to the clinical aspect of this study, there will be correlative studies where molecular response will be checked and its correlation with clinical response.

ELIGIBILITY:
Inclusion Criteria:

* WHO 2008 diagnosis of Polycythemia Vera Hemoglobin > 18.5 g/dl for men (16.5 g/dl for women) and presence of JAK2V617F mutation and either bone marrow trilineage myeloproliferation or subnormal serum erythropoietin level Patients may be on active treatment (phlebotomy, aspirin) ECOG performance status 0,1,2,or 3 Adequate hepatic function, adequate renal function

Exclusion Criteria:

* Patient with active malignancy Patients with clinically significant cardiac disease within 1 year Opthalmologic or gastrointestinal abnormalities Concurrent cytoreductive therapy is not allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Cherry, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: we conducted a single arm, prospective phase II study at the University of Oklahoma Health Sciences Center and the Oklahoma City VA hospitals in patients withWHO-defined JAK2V617F-positive PV from June 2010 to August 2012
Pre-assignment Details: Patients were eligible for the study if they were at least 18 years of age and had a diagnosis of PV per WHO 2008 criteria. Additional eligibility criteria included adequate liver and kidney function tests and an ECOG performance status of 0, 1, 2, or 3.
Period: Overall Study
Arm/Group | +JAK2V61F Mutation
Started | 5
Completed | 3
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: patients diagnosed with JAK2V617F-positive PV
Arm/Group | +JAK2V61F Mutation
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 63 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate to Include Complete Hematological Response, Complete Molecular Response, Partial Hematological Response, and Minimal Hematological Response
Time Frame: Day 15
Measure: Number; unit: participants
Groups:
- Single Arm Study: This was a single arm study
Arm/Group | Single Arm Study
Number analyzed (Participants) | 5
participants | 0

2. Secondary Outcome: Incidence of Toxicities
Description: Grade 3 or grade 4 toxicities as measured by CTCAE v3.0
Time Frame: First assessment at day 15, subsequent assessments at 28 day intervals for an average of 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Erlotinib: 150 mg po daily x 16 weeks
Arm/Group | Erlotinib
Number analyzed (Participants) | 5
Participants | 5

3. Secondary Outcome: Improvement in Splenomegaly Size
Time Frame: 4 months, end of treatment and 12 months end of treatment
Population: no improvement in spleen size
Measure: Count of Participants; unit: Participants
Arm/Group | +JAK2V61F Mutation
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Decrease of Mutant JAK2V617F Allele Burden
Time Frame: every 2 months until end of treatment and 12 months after end of treatment
Population: did not achieve hematological response
Measure: Count of Participants; unit: Participants
Arm/Group | +JAK2V61F Mutation
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Arm/Group | +JAK2V61F Mutation
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | +JAK2V61F Mutation (N=5)
grade 3 colitis (Gastrointestinal disorders) | 1 (1)
grade 2 facial rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | +JAK2V61F Mutation (N=5)
Grade 1-2 Diarrhea (Gastrointestinal disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No